CLINICAL TRIAL: NCT01758926
Title: Association Between Inflammatory Activities and Epithelial Gap Density in Inflammatory Bowel Disease
Brief Title: Association Between Inflammatory Activities and Gap Density
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Chief of the Department of Gastroenterology, Qilu Hospital, Shandong University, Shandong University
Other Study IDs: 2012SDU-QILU-G03
Record Dates: First submitted 2012-12-27; First posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-12

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease; Confocal Laser Endomicroscopy
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Observational Study Model: Case-Control
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Inflammatory bowel disease: Patients previously diagnosed as having IBD
- Health control: Asymptomatic individuals admitted for health surveillance or patients for follow up after polypectomy.

SUMMARY:
The study aims to:

1. To determine the relationship between inflammatory activities and epithelial gaps in IBD by CLE and evaluate epithelial gaps healing via dexamethasone treatment.
2. To demonstrated the alteration of local barrier function in IBD using CLE.

DETAILED DESCRIPTION:
The primary end-point of this study was the cohort comparison of epithelial gap density and local barrier function as determined by CLE of subjects with IBD versus controls. Despite discontinuities in the cellular layer, the intestinal barrier function is maintained during this high cell turnover rate at the apical pole of the epithelial layer. Gaps first identified in vivo through acriflavine have pivotal definitions (lacked nuclei or cytosol, appeared to be filled with an impermeable substance). However, Current endoscopic technology does not identify whether there is material present in human gaps, so investigators could not formally resolve whether human epithelial gaps compromise or defend the epithelial barrier.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 18-80
* IBD： Patients previously diagnosed as having IBD
* Health control: Asymptomatic individuals admitted for health surveillance or patients for follow up after polypectomy.
* Subjects who experienced successful intubation of the terminal ileum.

Exclusion Criteria:

* Subjects age < 18 or >80 years
* Subjects under conditions unsuitable for performing CLE including coagulopathy (prothrombin time <50% of control, partial thromboplastin time >50 s), cirrhosis, renal dysfunction (creatinine level >1.2 mg/dL), pregnancy or breastfeeding, acute gastrointestinal bleeding, jaundice and known allergy to fluorescein sodium.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with indications for colonoscopy in Qilu Hospital outpatient and inpatient department.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
gap density | 6 months
  the distributions of gap density

SECONDARY OUTCOMES:
local barrier function | 6 months
  the comparison local barrier function between the IBD group and normal control patients

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD, PhD, Study Director — Department of Gastroenterology, Qilu Hospital
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China